CLINICAL TRIAL: NCT01393366
Title: Facing Obstacles to RDI(Relative Dose Intensity)Through Telephone Intervention Strategy
Brief Title: Facing Obstacles to RDI (Relative Dose Intensity) Through Telephone Intervention Strategy
Acronym: FORTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1030903
Record Dates: First submitted 2011-07-05; First posted 2011-07-13 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without AMA (Other): Patient will be follow only like usual practice
  Interventions: Other: Usual Practice
- With AMA (Other): Patient will be follow like usual practice, plus 'Telephone Intervention' every week with a nurse to evaluate physical conditions.
  Interventions: Other: Telephone Intervention

INTERVENTIONS:
Other: Telephone Intervention — Only for arm AMA, patient will have one phone every week to evaluate physical conditions.
  Arms: With AMA
Other: Usual Practice — None, only usual practice.
  Arms: Without AMA

SUMMARY:
The investigators plan to conduct a nurse-based telephone intervention study to minimize toxicity and increase compliance to a combination of Fludarabine-Cyclophosphamide-Rituximab (FCR) given frontline to Chronic Lymphocytic Leukemia patients.

ELIGIBILITY:
Inclusion Criteria:

1. CLL whatever Binet stage, but with at least one NCIWG2008 criteria indicating a need for first line treatment.

   * Matutes score must be 4-5/5.
   * Initial cytopenia (due to CLL) are not exclusion criteria.
   * Lymph node biopsy is needed only if suspicion of Richter syndrome.
   * Mandatory pre-therapeutic check-up: FISH in search for deletion del17p and del11q, DAT test, haptoglobin levels, creatinine clearance.
2. Eligibility to a treatment with FCR: clearance > 60ml/mn, consider dose adjustments (recommended by protocol) if clearance30-60ml/mn, and comorbidity score CIRS-G≤11.
3. Signed informed consent
4. Age> or equal 18 years, ECOG PS 0-2.
5. Estimated overall survival>6 months.
6. Conserved liver function (bilirubin<2,5mg/dl, SGPT<4ULN, SGOT<4ULN) except infiltration due to the disease.
7. Contraception for younger patients.
8. Confident with the use of telephone, no disabling deafness.

Exclusion Criteria:

1. Richter syndrome or atypical CLL (Matutes score <4), and/or del17p by FISH
2. Relapse of CLL
3. Contra-indications to fludarabine: auto-immune cytopenia, creatinine clearance<30 ml/mn.
4. Serologies positive for HIV, HBV, or HCV. No active bacterial, viral or fungal infection
5. Previous history of hypersensibility to any product used in this protocol
6. Denial, or medical or psychological condition preventing completion of the signed informed consent.
7. Treatment with an investigational agent, or participation to another therapeutic protocol, 30 days before participating to this study.
8. Pregnant/breastfeeding women.
9. CNS involvement by CLL.
10. Presence of another cancer needing treatment (except basocellular carcinoma or cervix cancer managed with only surgery or local therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of RDI | 3 years
  Reductions in Relative Dose Intensity, calculated as the difference between initially planned doses of F, C and R and effectively prescribed doses of the 3 drugs, before and after 6 courses of FCR.

SECONDARY OUTCOMES:
Evaluation of Toxicity grade III-IV | 3 years
  rate of grade III-IV toxicities (neutropenia, fever, infections, renal insufficiency), assessment of quality of life and psychological comfort during FCR therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Loïc YSEBAERT, MD, Principal Investigator — University Hospital Of Toulouse
Locations (3):
- France (3):
  - Centre Hospitalier de la côte basque, Bayonne
  - CH Saint Jean, Perpignan
  - CHU Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ysebaert L, Larcher M, Compaci G, Oberic L, Sahnes L, Banos A, Araujo C, Sommet A, Laurent G, Despas F. Oncology nurse phone calls halve the risk of reduced dose intensity of immunochemotherapy: results of the randomized FORTIS study in chronic lymphocytic leukemia. Ann Hematol. 2019 Apr;98(4):931-939. doi: 10.1007/s00277-019-03631-z. Epub 2019 Feb 18. PMID 30778715